CLINICAL TRIAL: NCT06187714
Title: Effect of Caudal Block Injection Rate on Optic Nerve Sheath Diameter in Pediatric Surgeries
Status: Completed | Type: Observational
Sponsor: Prof. Dr. Cemil Tascıoglu Education and Research Hospital Organization (Other)
Responsible Party: Principal Investigator, Rasim Onur Karaoglu, MD, Prof. Dr. Cemil Tascıoglu Education and Research Hospital Organization
Other Study IDs: 681429
Record Dates: First submitted 2023-12-17; First posted 2024-01-03 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2024-08

CONDITIONS: Optic Nerve Sheath Diameter; Caudal Block

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- 0.25ml/sec
  Interventions: Procedure: caudal block rate
- 0.5ml/sec dose
  Interventions: Procedure: caudal block rate

INTERVENTIONS:
Procedure: caudal block rate — optic nerve sheath diameter measurement according to caudal block rate

SUMMARY:
Our prospective observational study will include patients between the ages of 1-7 years, ASA 1-2, who will undergo elective surgery under general anesthesia, whose consent was obtained by their parents for the procedure to be performed. Optic nerve sheath diameter of the patients will be measured and recorded.

DETAILED DESCRIPTION:
The study will be conducted with patients who will undergo elective surgery and caudal block will be applied between 05.07.2023-05.09.2023 in the Anesthesiology and Reanimation Clinic of Prof. Dr. Cemil Taşçıoğlu City Hospital after Ethics Committee approval and written and verbal consent of the patients. Our prospective observational study will include patients between the ages of 1-7 years, ASA 1-2, who will undergo elective surgery under general anesthesia, whose consent was obtained by their parents for the procedure to be performed. Gender, age, weight, height, body mass index (BMI), ASA (American Society of Anesthesiology) score and medical history of the patients will be recorded. Injection times of pediatric patients who underwent caudal block with 0.125% bupivacaine at a dose of 0.8 ml/kg using a 22 gauge caudal needle will be noted. Optic nerve sheath diameter of the patients will be measured and recorded. Intraoperative hemodynamic parameters, postoperative complications (nausea, vomiting, urinary retention) will also be noted.

ELIGIBILITY:
Inclusion Criteria:

Patients aged 1-7 years, ASA 1-2, who will undergo elective surgery under general anesthesia, in whom consent has been obtained for the procedure to be performed

Exclusion Criteria:

-

Ages: 1 Year to 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: pediatric patients aged 1-7 years for caudal block
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2023-07-05 (Actual); Primary Completion 2023-10-05 (Actual); Study Completion 2024-02-05 (Actual)

PRIMARY OUTCOMES:
optic nerve sheath diameter measurement | 1st minute after caudal block
  optic nerve sheath diameter

SECONDARY OUTCOMES:
optic nerve sheath diameter measurement | 10th minute after caudal block
  optic nerve sheath diameter

OTHER OUTCOMES:
optic nerve sheath diameter measurement | 20th minute after caudal block
  optic nerve sheath diameter

CONTACTS AND LOCATIONS:
Locations (1):
- Prof. Dr. Cemil Tascioglu City Hospital, Istanbul, Sisli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF